CLINICAL TRIAL: NCT00271674
Title: YAG Laser Versus Punch Biopsy for the Treatment of Tattoo Skin Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KF-01-275533
Record Dates: First submitted 2006-01-03; First posted 2006-01-04 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-06

CONDITIONS: Tattoo Skin Markers

INTERVENTIONS:
Device: Q-switched YAG laser

SUMMARY:
The purpose of the study is to compare patient satisfaction, clinical efficacy and adverse effects of Q-switched YAG laser versus punch biopsies for the treatment of tattoo dots that are applied as skin markers in relation to X-ray treatment of malignant disorders.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* Skin types I-IV,
* No previous laser treatment for the condition.

Exclusion Criteria:

* Younger than 18 years,
* Skin types V-VI,
* Pregnant or lactating women,
* Previous laser treatment for the condition,
* Recent exposure to sun or sun-beds,
* Treatment with oral retinoids within 3 months,
* Tendency to produce hypertrophic scars or keloids,
* Immunosuppressive treatment or disorders

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2006-01; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merete Haedersdal, MD, PhD, DrMedSci., Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Copenhagen NV, Denmark